CLINICAL TRIAL: NCT01723202
Title: A Randomized Phase 2 Study of Single Agent Dabrafenib (BRAFi) vs. Combination Regimen Dabrafenib (BRAFi) and Trametinib (MEKi) in Patients With BRAF Mutated Thyroid Carcinoma
Brief Title: Dabrafenib With or Without Trametinib in Treating Patients With Advanced Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bhavana Konda (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, Bhavana Konda, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-12064; NCI-2012-01700 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCNGSK20008 (Other: National Comprehensive Cancer Network (NCCN))
Record Dates: First submitted 2012-10-22; First posted 2012-11-07 (Estimated); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Follicular Thyroid Cancer; Insular Thyroid Cancer; Papillary Thyroid Cancer; Recurrent Thyroid Cancer
Keywords: BRAF; BRAFi; thyroid cancer; thyroid carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: GSK2118436 (Experimental): Patients receive dabrafenib orally 2 twice a day on days 1-28. Patients with disease progression may cross over to arm II.
  Interventions: Drug: dabrafenib
- Arm B: GSK2118436 and GSK1120212 (Experimental): Patients receive dabrafenib orally twice a day and trametinib orally once a day on days 1-28.
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — 150 mg orally twice daily given orally
  Other Names: BRAF inhibitor GSK2118436; GSK2118436
Drug: trametinib — 150 mg orally twice daily and GSK1120212 (MEKi) 2 mg orally once daily given orally
  Other Names: GSK1120212; MEKi
  Arms: Arm B: GSK2118436 and GSK1120212

SUMMARY:
This randomized phase II trial studies how well dabrafenib works with or without trametinib in treating patients with recurrent thyroid cancer. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether dabrafenib is more effective when given with or without trametinib in treating thyroid cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To screen two different regimens (GSK2118436 [BRAFi] [dabrafenib] as a single agent versus the combination regimen of GSK2118436 [BRAFi] and GSK1120212 [MEKi] [trametinib]) and identify which regimen is more promising for subsequent testing in a phase III trial in radioiodine refractory BRAF-mutated differentiated thyroid cancer (DTC) patients.

SECONDARY OBJECTIVES:

I. To understand duration of objective response, progression-free survival and overall survival for each treatment group.

II. To assess tolerability and adverse events of GSK2118436 (BRAFi) as a single agent and the tolerability and adverse events of GSK2118436 (BRAFi) and GSK1120212 (MEKi) in combination, in patients with DTC.

III. To evaluate impact of experimental drugs on serum tumor marker thyroglobulin and its correlation with overall response rate.

IV. To understand pharmacokinetic, pharmacogenetics and pharmacodynamics of experimental drugs using serial tumor biopsies, tumor blocks and peripheral blood.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dabrafenib orally (PO) twice daily (BID) on days 1-28. Patients with disease progression may cross-over to arm II.

ARM II: Patients receive dabrafenib PO BID and trametinib PO once daily (QD) on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary thyroid cancer, follicular thyroid cancer (tall cell variant, insular thyroid cancer, follicular variant of papillary thyroid cancers, poorly differentiated thyroid cancer or any of the above mixed histology will be allowed)
* Presence of BRAF mutation in tumor tissue
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; malignant lymph nodes will be considered measurable if they are >= 15 mm in short axis
* Patients must have progressive disease within the thirteen months prior to study entry; progressive disease is as defined in Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, which is at least a 20% increase in the sum of diameters of target lesions and the sum must also demonstrate an absolute increase of at least 5 mm; the appearance of one or more new lesions is also considered progressive disease
* Patients are willing to have tumor biopsy pre-study and at 4 weeks on study (fine needle aspiration or core biopsy) if patient has biopsy-accessible tumors as determined by investigator
* Patients must have disease that is refractory (unresponsive) to radioactive iodine (RAI) treatment as defined by one of the following:

  * One or more measurable lesions that do not demonstrate RAI uptake
  * One or more measurable lesions progressive by RECIST 1.1 within 12-months of prior RAI therapy
  * Cumulative RAI dose of > 600 mCi
* Prior therapy allowed:

  * Patients may have been previously treated with up to three regimens of oral multikinase inhibitors, including sorafenib, sunitinib and pazopanib
  * Patients may have been previously treated with external beam radiation or cytotoxic chemotherapy therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Serum creatinine =< 1.5 X institutional upper limit of normal
* Left ventricular ejection fraction (EF) >= institutional lower limit of normal
* Patient must have a calcium phosphate product (CPP) =< 4.0 mmol^2/L^2 (50 mg^2/dL^2)
* Female patients of childbearing age are required to have a negative serum pregnancy test within 14 days prior to the first dose of study medication

  * Females are required to use an effective method of contraception from the time of negative serum pregnancy test, throughout the study duration, and until 4 weeks after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 16 weeks after completion of the last dose of study drug
  * Specific contraception requirements for females: female subjects of childbearing potential must not become pregnant and are required to be sexually inactive by abstinence or use contraceptive methods with a failure rate of < 1%; sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject; periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception; contraceptive methods with a failure rate of < 1% include the following:

    * Intrauterine device (IUD) or intrauterine system (IUS) that meets the < 1% failure rate as stated in the product label
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is patient's sole sexual partner; for this definition, "documented" refers to the outcome of the investigator's/qualified physician designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
    * Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository); these allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label; the investigator is responsible for ensuring subjects understand how to properly use these methods of contraception
  * Specific contraception requirements for males: to prevent pregnancy in a female partner or to prevent exposure of any partner to the investigational product from a male subject's semen, male subjects must use one of the following contraceptive methods during the study and for a total of 16 weeks following the last dose of study drug (based upon the lifecycle of sperm):

    * Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject for 14 days prior to first dose of study drug, through the dosing period, and for at least 16 weeks after the last dose of study drug; periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Condom (during non-vaginal intercourse with any partner - male or female) OR
    * Condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) (during sexual intercourse with a female)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients had external beam radiotherapy, cytotoxic chemotherapy, or oral multikinase inhibitors within 4 weeks prior to entering the study
* Patients who have been treated with radioactive iodine within 24 weeks prior to entering the study (radioactive iodine within 4 weeks will be allowed if negative post-treatment scan)
* Patients have not recovered from adverse events related to prior chemotherapy, radiation therapy or multikinase inhibitors to Common Terminology Criteria for Adverse Events (CTCAE) 4.0 grade 1 or less except for alopecia
* Patients have been previously treated with potent BRAF inhibitor or MEK inhibitor, including PLX4032/vemurafenib, ARQ 736; previous treatment with sorafenib is permitted
* Patients are receiving any other investigational agents
* Patients are on any medication that is on the list of prohibitive medications; patients on therapeutic dose of warfarin; this is due to potential for significant interactions between warfarin and study agents
* Patients with a known history of infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Patients with a history of other malignancy; patients who have been disease-free from other malignancy for 5 years or greater, or patients with a history of resected non-melanoma skin cancer, or patients with a history of treated in situ carcinoma will be allowed
* Patients with uncontrolled brain metastases; patients who are on a stable dose of corticosteroids for more than 1 month or off corticosteroids for 2 weeks can be enrolled; enzyme-inducing anti-epileptic drugs are not permitted
* Patients with a known history of retinal vein occlusion or central serous retinopathy, or predisposing factors to retinal vein occlusion (RVO) or central serous retinopathy (CSR) (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
* Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:

  * Evidence of new optic disc cupping
  * Evidence of new visual field defects
  * Intraocular pressure > 21 mm Hg as measured by tonography
* Patients with a known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients with class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system

  * Abnormal cardiac valve morphology (subjects with minimal abnormalities, can be entered on study with approval)
* Corrected QT (QTc) interval greater than or equal to 480 msecs (>= 500 msec for subjects with bundle branch block)
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women and nursing women are excluded from this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Subjects with a history of pneumonitis or interstitial lung disease
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 6 months
* History of uncontrolled arrhythmias; subjects with controlled atrial fibrillation for > 1 month prior to study day 1 are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Konda, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Harvard Medical School, Boston, Massachusetts
  - Ohio State University Medical Center, Columbus, Ohio
  - The University of Texas-MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Busaidy NL, Konda B, Wei L, Wirth LJ, Devine C, Daniels GA, DeSouza JA, Poi M, Seligson ND, Cabanillas ME, Sipos JA, Ringel MD, Eisfeld AK, Timmers C, Shah MH. Dabrafenib Versus Dabrafenib + Trametinib in BRAF-Mutated Radioactive Iodine Refractory Differentiated Thyroid Cancer: Results of a Randomized, Phase 2, Open-Label Multicenter Trial. Thyroid. 2022 Oct;32(10):1184-1192. doi: 10.1089/thy.2022.0115. Epub 2022 Jul 5. PMID 35658604
- [Derived] Hicks HM, Pozdeyev N, Sams SB, Pugazhenthi U, Bales ES, Hofmann MC, McKenna LR, Schweppe RE. Fibronectin Contributes to a BRAF Inhibitor-driven Invasive Phenotype in Thyroid Cancer through EGR1, Which Can Be Blocked by Inhibition of ERK1/2. Mol Cancer Res. 2023 Sep 1;21(9):867-880. doi: 10.1158/1541-7786.MCR-22-1031. PMID 37219859
- [Derived] Owen DH, Konda B, Sipos J, Liu T, Webb A, Ringel MD, Timmers CD, Shah MH. KRAS G12V Mutation in Acquired Resistance to Combined BRAF and MEK Inhibition in Papillary Thyroid Cancer. J Natl Compr Canc Netw. 2019 May 1;17(5):409-413. doi: 10.6004/jnccn.2019.7292. PMID 31085763
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Dabrafenib Alone: Patients receive dabrafenib orally 2 twice a day on days 1-28. Patients with disease progression may cross over to arm II.
  dabrafenib: 150 mg orally twice daily given orally
  Correlative Studies: 1. Signaling inhibition studies in tumor biopsies (10 pts in each arm; 5 pts per center) 2. BRAF mutation studies in circulating plasma DNA (all study patients) 3. Mechanisms of drug resistance in tumor biopsies or tumor blocks (5 pts in each arm) 4. Assess predictors of response (Archival tumor block/unstained slides in all study patients) 5. Pharmacokinetic studies (First 10 pts enrolled on each arm) 6. Pharmacogenomics studies (All study patients)
- Arm B: Dabrafenib + Trametinib: Patients receive dabrafenib orally twice a day and trametinib orally once a day on days 1-28.
  dabrafenib: 150 mg orally twice daily given orally
  trametinib: 150 mg orally twice daily and GSK1120212 (MEKi) 2 mg orally once daily given orally
  Correlative Studies: 1. Signaling inhibition studies in tumor biopsies (10 pts in each arm; 5 pts per center) 2. BRAF mutation studies in circulating plasma DNA (all study patients) 3. Mechanisms of drug resistance in tumor biopsies or tumor blocks (5 pts in each arm) 4. Assess predictors of response (Archival tumor block/unstained slides in all study patients) 5. Pharmacokinetic studies (First 10 pts enrolled on each arm) 6. Pharmacogenomics studies (All study patients)
Period: Pre-crossover
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib
Started | 26 | 27
Completed | 26 | 27
Not Completed | 0 | 0
Period: Post-Crossover of Arm A Patients
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib
Started | 26 | 27
Dabrafenib Alone | 12 | 0
Dabrafenib + Trametinib | 14 | 27
Completed | 26 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dabrafenib Alone: Patients receive dabrafenib orally 2 twice a day on days 1-28. Patients with disease progression may cross over to arm II.
  dabrafenib: 150 mg orally twice daily given orally
  Correlative Studies: 1. Signaling inhibition studies in tumor biopsies (10 pts in each arm; 5 pts per center) 2. BRAF mutation studies in circulating plasma DNA (all study patients) 3. Mechanisms of drug resistance in tumor biopsies or tumor blocks (5 pts in each arm) 4. Assess predictors of response (Archival tumor block/unstained slides in all study patients) 5. Pharmacokinetic studies (First 10 pts enrolled on each arm) 6. Pharmacogenomics studies (All study patients)
- Dabrafenib + Trametinib: Patients receive dabrafenib orally twice a day and trametinib orally once a day on days 1-28.
  dabrafenib: 150 mg orally twice daily given orally
  trametinib: 150 mg orally twice daily and GSK1120212 (MEKi) 2 mg orally once daily given orally
  Correlative Studies: 1. Signaling inhibition studies in tumor biopsies (10 pts in each arm; 5 pts per center) 2. BRAF mutation studies in circulating plasma DNA (all study patients) 3. Mechanisms of drug resistance in tumor biopsies or tumor blocks (5 pts in each arm) 4. Assess predictors of response (Archival tumor block/unstained slides in all study patients) 5. Pharmacokinetic studies (First 10 pts enrolled on each arm) 6. Pharmacogenomics studies (All study patients)
- Total: Total of all reporting groups
Arm/Group | Dabrafenib Alone | Dabrafenib + Trametinib | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 84] | 65 [43 to 84] | 62.5 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate, Defined as the Proportion of Patients Who Have a Minor Response (MR), Partial Response (PR), or Complete Response(CR)Assessed According to RECIST.
Description: The MR+PR+CR response rate will be estimated for each treatment arm. In determining this rate, the number of patients with RECIST-based MR, PR or CR will be divided by the number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true PR+CR response rate will be calculated.
Time Frame: up to 24 weeks
Population: Participants were analyzed for objective response rate prior to the crossover of Arm A patients to Dabrafenib + Trametinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib
Number analyzed (Participants) | 26 | 27
percentage of participants | 42 [23 to 63] | 48 [29 to 68]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The MR+PR+CR response rate will be estimated for each treatment arm. In determining this rate, the number of patients with RECIST-based MR, PR or CR will be divided by the number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true PR+CR response rate
Time Frame: Up to 4 years or from start of treatment to time of progression or death
Measure: Median (Full Range); unit: months
Groups:
- Cross-over to Dabrafenib + Trametinib: Patients receive dabrafenib orally twice a day and trametinib orally once a day on days 1-28.
  dabrafenib: 150 mg orally twice daily given orally
  trametinib: 150 mg orally twice daily and GSK1120212 (MEKi) 2 mg orally once daily given orally
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib | Cross-over to Dabrafenib + Trametinib
Number analyzed (Participants) | 26 | 27 | 14
months | 10.7 [3.8 to 34.7] | 15.1 [12.3 to 37.3] | 7.5 [2.8 to 38.5]

3. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate overall survival. We will also evaluate the proportion of patients who are alive at one year.
Time Frame: up to 4 weeks after study treatment
Measure: Median (Full Range); unit: months
Arm/Group | Dabrafenib Alone | Dabrafenib + Trametinib | Cross-over to Dabrafenib + Trametinib
Number analyzed (Participants) | 26 | 27 | 14
months | 37.9 [23.4 to NA] — Upper limit not reached due to insufficient number of participants with events | 47.5 [27.9 to 57.8] | 36 [23.4 to NA] — Upper limit not reached due to insufficient number of participants with events

4. Secondary Outcome: Number of Adverse Events Related to Treatment With GSK2118436 (BRAFi) as a Single Agent and Adverse Events Related to Treatment With GSK2118436 (BRAFi) and GSK1120212 (MEKi) in Combination.
Description: Frequency and severity of adverse events in each of the treatment arms will be collected and summarized using descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The incidence of severe (grade 3+) adverse events or toxicities will be described.
Time Frame: Every 2 weeks for the first 8 weeks, and then every 4-8 weeks thereafter up to 4 weeks after completion of study treatment, up to 1 year
Measure: Number; unit: number of events
Groups:
- Crossover to Dabrafenib + Trametinib: Patients receive dabrafenib orally twice a day and trametinib orally once a day on days 1-28.
  dabrafenib: 150 mg orally twice daily given orally
  trametinib: 150 mg orally twice daily and GSK1120212 (MEKi) 2 mg orally once daily given orally
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib | Crossover to Dabrafenib + Trametinib
Number analyzed (Participants) | 26 | 27 | 14
number of events
  Anemia | 11 | 8 | 1
  Blood and lymphatic disorders- other | 1 | 4 | 0
  Sinus tachycardia | 1 | 0 | 0
  Hypothyroidism | 1 | 0 | 0
  Dry Eye | 1 | 1 | 1
  Eye disorders - other | 1 | 2 | 0
  Keratitis | 1 | 1 | 0
  Photophobia | 1 | 0 | 0
  Uveitis | 1 | 1 | 0
  Abdominal distension | 1 | 0 | 0
  Abdominal pain | 3 | 0 | 0
  Constipation | 1 | 1 | 0
  Diarrhea | 4 | 7 | 1
  Dry mouth | 1 | 1 | 0
  Dysphagia | 1 | 0 | 0
  Gastric hemorrhage | 1 | 0 | 0
  Gastric ulcer | 1 | 0 | 0
  Gastrointestinal disorders - other | 2 | 0 | 1
  Lower gastrointestinal hemorrhage | 1 | 0 | 0
  Nausea | 11 | 14 | 1
  Pancreatitis | 2 | 0 | 0
  Vomiting | 7 | 6 | 2
  Chills | 11 | 14 | 4
  Edema limbs | 3 | 5 | 1
  Fatigue | 10 | 14 | 1
  Fever | 13 | 16 | 6
  Flu like symptoms | 2 | 4 | 0
  Non-cardiac chest pain | 1 | 0 | 1
  Pain | 2 | 2 | 0
  Hepatobiliary disorders - other | 1 | 1 | 1
  Infections and infestations - other | 1 | 1 | 0
  Dermatitis radiation | 1 | 0 | 0
  Aspartate aminotransferase increased | 2 | 10 | 0
  Blood bilirubin increased | 1 | 0 | 0
  Creatinine increased | 1 | 2 | 0
  Ejection fraction decreased | 3 | 1 | 2
  Electrocardiogram QT corrected interval prolonged | 1 | 3 | 0
  Investigations - other | 2 | 4 | 2
  Lipase increased | 2 | 0 | 0
  Lymphocyte count decreased | 5 | 4 | 3
  Platelet count decreased | 3 | 2 | 0
  Weight loss | 7 | 2 | 0
  White blood cell decreased | 2 | 2 | 0
  Anorexia | 6 | 9 | 3
  Hyperglycemia | 12 | 5 | 5
  Hyperkalemia | 2 | 0 | 0
  Hypertriglyceridemia | 1 | 0 | 0
  Hypoalbuminemia | 2 | 2 | 1
  Hypokalemia | 1 | 1 | 0
  Hyponatremia | 2 | 1 | 0
  Hypophosphatemia | 9 | 11 | 3
  Metabolism and nutrition disorders - other | 1 | 3 | 1
  Arthralgia | 6 | 3 | 1
  Arthritis | 2 | 0 | 0
  Back pain | 1 | 0 | 0
  Bone pain | 1 | 1 | 0
  Generalized muscle weakness | 1 | 5 | 1
  Muscle weakness upper limb | 1 | 0 | 0
  Musculoskeletal and connective tissue disorder - Other | 1 | 2 | 0
  Myalgia | 5 | 6 | 0
  Neck pain | 1 | 0 | 0
  Pain in extremity | 1 | 0 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other | 3 | 0 | 0
  Concentration impairment | 1 | 0 | 1
  Dizziness | 3 | 1 | 0
  Dysgeusia | 1 | 1 | 0
  Encephalopathy | 1 | 0 | 0
  Headache | 5 | 3 | 1
  Nervous system disorders - Other | 1 | 0 | 0
  Anxiety | 1 | 0 | 0
  Confusion | 1 | 1 | 0
  Urinary frequency | 1 | 0 | 0
  Reproductive system and breast disorders - Other | 1 | 0 | 0
  Cough | 2 | 1 | 1
  Dyspnea | 1 | 2 | 1
  Hoarseness | 2 | 1 | 1
  Productive cough | 1 | 0 | 0
  Sore throat | 1 | 0 | 0
  Alopecia | 11 | 2 | 3
  Dry skin | 1 | 0 | 1
  Nail ridging | 1 | 0 | 1
  Palmar-plantar erythrodysesthesia syndrome | 11 | 6 | 4
  Photosensitivity | 1 | 0 | 0
  Pruritus | 6 | 3 | 0
  Rash maculo-papular | 7 | 4 | 2
  Scalp pain | 1 | 0 | 0
  Skin and subcutaneous tissue disorders - Other | 17 | 9 | 2
  Flushing | 1 | 0 | 0
  Hot flashes | 1 | 0 | 0
  Hypertension | 2 | 4 | 1
  Hypotension | 1 | 0 | 0
  Aortic valve disease | 0 | 1 | 0
  Cardiac disorders - Other | 0 | 1 | 1
  Blurred vision | 0 | 4 | 0
  Floaters | 0 | 1 | 0
  Retinal vascular disorder | 0 | 1 | 0
  Colonic hemorrhage | 0 | 1 | 0
  Duodenal hemorrhage | 0 | 1 | 0
  Duodenal ulcer | 0 | 1 | 0
  Gastroesophageal reflux disease | 0 | 1 | 0
  Mucositis oral | 0 | 3 | 0
  General disorders and administration site conditions - Other | 0 | 3 | 0
  Irritability | 0 | 1 | 0
  Cholecysitis | 0 | 1 | 0
  Papulopustular rash | 0 | 3 | 0
  Fall | 0 | 1 | 0
  Alanine aminotransferase increased | 0 | 8 | 0
  Alkaline phosphatase increased | 0 | 5 | 0
  Neutrophil count decreased | 0 | 3 | 0
  Hypercalcemia | 0 | 1 | 0
  Hypocalcemia | 0 | 3 | 0
  Chest wall pain | 0 | 1 | 0
  Depressed level of consciousness | 0 | 1 | 0
  Memory impairment | 0 | 2 | 0
  Paresthesia | 0 | 1 | 0
  Peripheral sensory neuropathy | 0 | 1 | 0
  Seizure | 0 | 1 | 0
  Spasticity | 0 | 1 | 0
  Urinary incontinence | 0 | 1 | 0
  Dysmenorrhea | 0 | 1 | 0
  Epistaxis | 0 | 2 | 0
  Erythema multiforme | 0 | 1 | 0
  Rash acneiform | 0 | 1 | 1
  Telangiectasia | 0 | 1 | 0
  Urticaria | 0 | 1 | 0
  Thromboembolic even | 0 | 1 | 0
  Thrombotic thrombocytopenic purpura | 0 | 1 | 1
  Left ventricular systolic dysfunction | 0 | 1 | 1
  Psychiatric disorders - Other | 0 | 0 | 1

5. Secondary Outcome: Tolerability of the Regimens in Terms of the Number of Patients Who Required Dose Modifications and/or Dose Delays.
Description: Tolerability of the regimen in each of the treatment arms will be collected and summarized using descriptive statistics. We will also capture the proportion of patients who go off treatment due to adverse reactions or even those who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial. These tolerability measures will be assessed within each of the treatment arms and we will explore differences in these measures between the arms.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib | Cross-over to Dabrafenib + Trametinib
Number analyzed (Participants) | 26 | 27 | 14
Participants
  Dose Reductions | 6 | 15 | 4
  Permanent Discontinuations | 5 | 6 | 2

ADVERSE EVENTS:
Time Frame: The severity of adverse events will be graded utilizing the National Cancer Institutes Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) up to 1 year. All-Cause Mortality was assessed up to 5 years.
Arm/Group | Arm A: Dabrafenib Alone | Arm B: Dabrafenib + Trametinib | Crossover to Dabrafenib + Trametinib
All-Cause Mortality (participants affected / at risk) | 9/26 | 8/27 | 2/14
Serious Adverse Events (participants affected / at risk) | 6/26 | 6/27 | 0/14
Other Adverse Events (participants affected / at risk) | 26/26 | 27/27 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Dabrafenib Alone (N=26) | Arm B: Dabrafenib + Trametinib (N=27) | Crossover to Dabrafenib + Trametinib (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | NA
Dysphagia (Nervous system disorders) | 1 (1) | 0 (0) | NA
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Fatigue (General disorders) | 1 (1) | 0 (0) | NA
Papillary urothelial carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | NA
Fever (General disorders) | 0 (0) | 4 (6) | NA
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1) | NA — possible cardiac ischemia
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1) | NA
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Chills (General disorders) | 0 (0) | 1 (1) | NA
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | NA
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | NA
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | NA
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Dabrafenib Alone (N=26) | Arm B: Dabrafenib + Trametinib (N=27) | Crossover to Dabrafenib + Trametinib (N=14)
Anemia (Blood and lymphatic system disorders) | 17 (17) | 16 (16) | 4 (4)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Hypothyrodism (Endocrine disorders) | 4 (4) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Eye disorders - Other (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (7) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 11 (11) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (14) | 17 (17) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10) | 8 (8) | 2 (2)
Chills (General disorders) | 11 (11) | 16 (16) | 4 (4)
Edema limbs (General disorders) | 6 (6) | 9 (9) | 5 (5)
Fatigue (General disorders) | 16 (16) | 21 (21) | 6 (6)
Fever (General disorders) | 14 (14) | 17 (17) | 6 (6)
Flu like symptoms (General disorders) | 3 (3) | 9 (9) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 5 (5) | 8 (8) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2) | 2 (2)
Pain (General disorders) | 9 (9) | 5 (5) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4) | 7 (7) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 8 (8) | 0 (0)
Alkaline phosphatase increased (Investigations) | 10 (10) | 11 (11) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 15 (15) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 4 (4) | 6 (6) | 2 (2)
Ejection fraction decreased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (3) | 5 (5) | 1 (1)
Investigations - Other (Investigations) | 9 (9) | 7 (7) | 5 (5)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (11) | 10 (10) | 8 (8)
Platelet count decreased (Investigations) | 4 (4) | 6 (6) | 0 (0)
Weight gain (Investigations) | 2 (2) | 6 (6) | 1 (1)
Weight loss (Investigations) | 11 (11) | 5 (5) | 3 (3)
White blood cell decreased (Investigations) | 4 (4) | 5 (5) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 15 (15) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (22) | 20 (20) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 9 (9) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 11 (11) | 9 (9) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (11) | 13 (13) | 3 (3)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 6 (6) | 3 (3)
Nervous system disorders - Other (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 12 (12) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (14) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 2 (2) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (11) | 8 (8) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (6) | 4 (4)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 19 (19) | 11 (11) | 4 (4)
Hot flashes (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 15 (15) | 13 (13) | 7 (7)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Vascular disorders, other (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac Disorders- other (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 5 (5) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT01723202/Prot_SAP_000.pdf